CLINICAL TRIAL: NCT00009191
Title: The Depression in Alzheimer's Disease Study (DIADS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH056511 (NIH); R01MH056511 (NIH); IA0010; DSIR AT-GP; NCT00000182 (obsolete NCT alias)
Record Dates: First submitted 2001-01-23; First posted 2001-01-24 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer Disease; Depression
MeSH Terms: conditions — Alzheimer Disease; Depression | interventions — Sertraline

INTERVENTIONS:
Drug: Sertraline [Zoloft]

SUMMARY:
Major depression afflicts approximately 25 percent of patients with AD. Depression in AD patients leads to mental suffering, behavioral disturbance (such as aggression), poor cognition, poor self-care, caregiver depression, caregiver burden, and early entry into the nursing home. Since major depression is treatable, this additional disability may be avoidable. The use of antidepressants to treat major depression in AD is supported by two studies, although a third does not show a benefit for antidepressants over placebo. Also, the safety of antidepressant treatment in depressed AD patients is poorly studied. A conclusive study showing that depression reduction in AD can be accomplished safely with antidepressant medications, and that depression reduction is associated with improvements in activities of daily living, non-mood behavioral disturbances, caregiver burden, and caregiver depression would have major clinical and cost implications for the care of the AD patient. This study is a 13-week, double blind, flexible dose, placebo controlled trial of sertraline in the treatment of outpatients with AD and co-morbid major depression. The hypothesis is that antidepressant treatment is superior to placebo in improving mood, in improving cognition, in reducing physical dependency, in reducing caregiver depression, and in reducing caregiver burden. It is also hypothesized that the degree of depression reduction is correlated with these improvements. It is further hypothesized that the safety profile of sertraline when compared to placebo is acceptable, especially with regard to risk of falls, sleep disturbance, and delirium. One hundred community residing outpatients with probable AD who also meet DSM-IV criteria for major depressive episode will be recruited into the study. They will be randomized to sertraline or placebo and followed through weekly telephone contact by an experienced clinical trials team. Outcomes will be assessed every 3 weeks, for a total of four followup data points. Scales assessing the following domains will be used: depression, cognition, behavioral disturbance, physical dependency, delirium, falls, sleep, other side effects, caregiver depression, caregiver burden, caregiver functioning, and caregiver health.

ELIGIBILITY:
Inclusion:

* Diagnosis of Probable Alzheimer's disease (AD) by NINCDS/ADRDA criteria (McKann et al., 1984), with a MMSE score greater than 10
* Diagnosis of current major depressive episode (MD), by DSM-IV, based on the SCID-IV examination
* Patients will be included even if they have a pre-AD history of unipolar depression
* Patients who currently are being treated with antidepressants but continue to meet criteria for MD (i.e., have not responded to the medications) and who are willing to discontinue the other medication and enter the study also will be included
* Currently residing in the community (own home,family member's home, or small group home) and agreeing to 13 weeks of followup in the study
* Stable medical history and general health, in the opinion of the study psychiatrist
* A caregiver who knows the patient well (spends at least 10 hours per week with him or her), and who is in reasonably good health, agrees to participate as well
* Participant and his/her legal representative provide informed consent

Exclusion:

* Use of sertraline is contraindicated, based on the Food and Drug Administration package insert for sertraline
* Patient has a lifetime diagnosis of schizophrenia, bipolar disorder, or pre-AD anxiety disorder, as determined by the SCID
* Patient has a current substance use disorder, as determined by the SCID
* Patient is acutely suicidal or requires inpatient psychiatric hospitalization, as determined by the study psychiatrist
* No psychotropic medicine dose changes, including cholinesterase inhibitors, after study entry
* May enter with any drug except another antidepressant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-11; Primary Completion 2006-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Lyketsos CG, Sheppard JM, Steele CD, Kopunek S, Steinberg M, Baker AS, Brandt J, Rabins PV. Randomized, placebo-controlled, double-blind clinical trial of sertraline in the treatment of depression complicating Alzheimer's disease: initial results from the Depression in Alzheimer's Disease study. Am J Psychiatry. 2000 Oct;157(10):1686-9. doi: 10.1176/appi.ajp.157.10.1686. PMID 11007727